CLINICAL TRIAL: NCT00930553
Title: An Extension Protocol for Multiple Sclerosis Patients Who Participated in Genzyme-Sponsored Studies of Alemtuzumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAMMS03409; 2009-010788-18 (EudraCT Number); LTE12824 (Other: Sanofi)
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Previously treated with alemtuzumab (Experimental): Alemtuzumab 12 mg per day administered through IV, once a day for 3 consecutive days (participants might receive additional cycles of alemtuzumab upon documented evidence of resumed disease activity, but not within same 12-month period)
  Interventions: Biological: alemtuzumab
- Previously treated with interferon beta-1a (Rebif®) (Experimental): Alemtuzumab 12 mg per day administered through IV, once a day for 5 consecutive days during the first cycle and 12 mg per day administered through IV, once a day for 3 consecutive days during the second cycle, 12 months later. Participants might qualify for as-needed retreatment (12 mg per day administered through IV, once a day for 3 consecutive days) after their second fixed annual cycle.
  Interventions: Biological: alemtuzumab

INTERVENTIONS:
Biological: alemtuzumab — Alemtuzumab 12 mg/day IV infusion on 5 consecutive days if the participants had no prior alemtuzumab exposure (ie, first treatment course). All subsequent treatment courses were for 3 days only.

SUMMARY:
This open-label, rater-blinded extension study enrolled participants who had relapsing-remitting multiple sclerosis (RRMS) and who participated in one of three prior Genzyme-sponsored studies of alemtuzumab (CAMMS223 [NCT00050778], CAMMS323 [NCT00530348] also known as CARE-MS I, or CAMMS324 [NCT00548405] also known as CARE-MS II). The purposes of this study were:

1. To examine the long term safety and efficacy of alemtuzumab treatment in participants who received alemtuzumab as their study treatment in one of the prior studies.
2. To examine the safety and efficacy of initial alemtuzumab treatment in this study for participants who received Rebif® (interferon beta-1a) as their study treatment in one of the prior studies.
3. To determine the safety and efficacy of additional "as needed" alemtuzumab treatment courses. This applied both to participants who received alemtuzumab for the first time in one of the prior studies or for the first time in this extension study.

DETAILED DESCRIPTION:
Alemtuzumab treatment was on a fixed schedule of two treatment courses a year apart for participants who received Rebif® in one of the prior Genzyme-sponsored studies of alemtuzumab or on an as needed schedule (e.g. due to documented evidence of resumed Multiple Sclerosis [MS] activity) for participants who had already completed a fixed schedule of treatment with alemtuzumab in one of the prior Genzyme-sponsored studies. There was no comparison treatment in this study. All participants were required to return to their study site every 3 months for neurologic and other assessments. In addition, safety-related laboratory tests and surveys were performed at least monthly. Participation in the extension study was at least 48 months from enrollment. Study duration could be extended to allow participants to remain in the study until a follow-up study was available in their country or through month 60 (month 72 in USA), whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* 1.Received alemtuzumab in CAMMS323 or CAMMS324, completed the 2-year study period, and had not subsequently received disease modifying treatments (other than glatiramer acetate or interferon beta); or
* 2.Received Rebif® in CAMMS323 or CAMMS324, completed the 2-year study period, and had not subsequently received alternative disease modifying treatments (other than glatiramer acetate or another interferon beta); or
* 3.Participated in CAMMS223.
* NOTE: Criteria 1 and 2 above meant that participants who enrolled in CAMMS323 or CAMMS324 but did not complete the 2-year study period or went on to receive non-study drug DMTs after randomization were not eligible for inclusion in the Extension Study. Participants who enrolled in CAMMS324 after participation in CAMMS223 must meet criteria 1 or 2 to be eligible for inclusion in the Extension Study.

Exclusion Criteria:

* Any alemtuzumab participant from CAMMS223, CAMMS323, or CAMMS324 who had received alemtuzumab off-label (ie, outside of one of the prior Genzyme-sponsored studies), or was participating in any other investigational study, unless approved by Genzyme. In addition, these participants must be screened for disqualifying safety concerns before receiving alemtuzumab retreatment.
* Any Rebif® participants from CAMMS223, CAMMS323, or CAMMS324 who met any of the following criteria. In addition, these participants must be screened for disqualifying safety concerns before receiving alemtuzumab treatment. a) Did not wish to receive alemtuzumab; b) Ongoing participation in any other investigational study, unless approved by Genzyme; c) Had received alemtuzumab off-label (ie, outside of one of the prior Genzyme-sponsored studies); d) Known bleeding disorder or therapeutic anticoagulation; e) Diagnosis of idiopathic thrombocytopenia purpura or other autoimmune hematologic abnormality; f) History of malignancy, except basal cell skin carcinoma; g) Intolerance of pulsed corticosteroids, especially a history of steroid psychosis h) Significant Autoimmune disorder (other than MS); i) Major psychiatric disorder or epileptic seizures not adequately controlled by treatment; j) Active infection or high risk for infection k) Unwilling to use a reliable and acceptable contraceptive method during and for at least 6 months following each alemtuzumab treatment cycle (fertile participants only).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1314 (Actual)
Dates: Start 2009-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme Coorporation
Locations (176):
- United States (69):
  - North Central Neurology Associates, P.C., Cullman, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center Barrow Neurology Clinics - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Arizona (Scottsdale), Scottsdale, Arizona
  - Northwest NeuroSpecialists, PLLC, Tucson, Arizona
  - East Bay Physicians Medical Group/ Sutter East Bay Medical Foundation, Berkeley, California
  - Neurology Center North Orange County, La Habra, California
  - University of Southern California Keck School of Medicine/University of Southern California LAC & USC Medical Center, Los Angeles, California
  - Neuro-Therapeutics, Inc., Pasadena, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Health Science Center - Aurora, Aurora, Colorado
  - Advanced Neurology of Colorado, Fort Collins, Colorado
  - Yale MS Research Center, New Haven, Connecticut
  - The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida Neuroscience Institute, Jacksonville, Florida
  - Neurology Associates, P.A., Maitland, Florida
  - Neurological Associates, Pompano Beach, Florida
  - Negroski, Stein, Sutherland and Hanes Neurology, Sarasota, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - Emory University Department of Neurology, Atlanta, Georgia
  - Shepherd Center Multiple Sclerosis Institute, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Consultants in Neurology, LTD, Northbrook, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Indiana University Multiple Sclerosis Center, Indianapolis, Indiana
  - Iowa Health Physicians, Des Moines, Iowa
  - Ruan Neurology Clinic and Clinical Research Center, Mercy Medical Center, Des Moines, Iowa
  - University of Kansas Medical Center, Department of Neurology, Kansas City, Kansas
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - Associates in Neurology, P.S.C., Lexington, Kentucky
  - Kentucky Neuroscience Research, Louisville, Kentucky
  - University of Maryland, Maryland Center for MS, Baltimore, Maryland
  - The MS Center at St. Elizabeth's, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Medical School, Ann Arbor, Michigan
  - Michigan Neurology Association, Clinton, Michigan
  - Wayne State University, The School of Medicine, Department of Neurology, Detroit, Michigan
  - Spectrum Health Medical Group, Neurology/Michigan Medical P.C., West Michigan MS Clinic, Grand Rapids, Michigan
  - Northern Michigan Neurology, Traverse City, Michigan
  - Saint Luke's Brain & Stroke Institute, Kansas City, Missouri
  - Renown Institute for Neurosciences, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - MS Center at Holy Name Hospital, Teaneck, New Jersey
  - University of New Mexico, Dept. of Neurology, Albuquerque, New Mexico
  - Empire Neurology P.C., Latham, New York
  - Winthrop University Hospital Multiple Sclerosis Treatment Center, Mineola, New York
  - MS Care Center at NYUMC and HJD, New York, New York
  - The Corinne Goldsmith Dickinson Center for Multiple Sclerosis at Mount Sinai, New York, New York
  - South Shore Neurologic Associates, P.C., Patchogue, New York
  - Rochester Multiple Sclerosis Center, Rochester, New York
  - SUNY Upstate Medical University, Department of Neurology, Syracuse, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Health Science Department of Neurology, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oak Clinic for Multiple Sclerosis, Uniontown, Ohio
  - OMRF Multiple Sclerosis Center of Excellence, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital Neurosciences and Pain Research, Allentown, Pennsylvania
  - Rhode Island Hospital MS Center - The Neurology Foundation, Inc, Providence, Rhode Island
  - Neurology Clinic PC, Cordova, Tennessee
  - Advanced Neurosciences Institute, Franklin, Tennessee
  - Hope Neurology, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Maxine Mesinger MS Clinic, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Integra Clinical Research, San Antonio, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - MS Center of Greater Washington, Vienna, Virginia
  - Swedish Medical MS Center, Seattle, Washington
- DIABAID, Buenos Aires, Argentina
- Australia (11):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Gold Coast Hospital, Southport, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - The Wesley Research Institute, Auchenflower QLD
  - The Queen Elizabeth Hospital, Woodville, SA
- AKH Wien-Universitätskliniken für Neurologie, Vienna, Austria
- Belgium (3):
  - Cliniques Universitaires Saint-luc, Brussels
  - CHU Ourthe Amblève, Esneux
  - University Hospital Leuven, Campus Gasthuisberg, Leuven
- Brazil (4):
  - Hospital Mae de Deus, Porto Alegre
  - Hospital da Restauração, Neurology department, Recife, PE
  - Irmandade da Santa Casa de Misericórdio de São Paulo, Neurology department, São Paulo, SP
  - Hospital das Clínicas da Faculdade de Medicina da USP, Neurology department, São Paulo,SP
- Canada (8):
  - University of Calgary, Department of Neurology, Calgary, Alberta
  - Kingston General Hospital MS Clinic, Kingston, Ontario
  - Clinique Neuro-Outaouais, Gatineau, Quebec
  - Recherche Sepmus, Inc., Greenfield Park, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - London Health Sciences Centre - University Hospital, London, on
  - The Ottawa Hospital - MS Research, Ottawa, Ontario
  - University of British Columbia, Vancouver, BC
- Croatia (6):
  - Clinical Hospital Osijek, Osijek
  - Clinical Hospital Centre Rijeka, Rijeka
  - General Hospital Varazdin, Department for Neurology, Varaždin
  - Clinical Hospital Centre "Sestre Milosrdnice", Zagreb
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Sveti Duh, Zagreb
- Czechia (4):
  - St. Anne's University Hospital Brno, Brno
  - University Hospital Hradec Králové, Hradec Králové
  - General Hospital, 128 21 Praha 2, Prague
  - Hospital Teplice, Neurology Department, MS centrum, Teplice
- Denmark (2):
  - Aarhus Sygehus, Århus C
  - Rigshospitalet Department of Neurology, Copenhagen
- France (5):
  - Hôpital Général, Dijon
  - Groupe Hospitalier Pitié-Salpêtrière, Fédération de Maladies du System Nerveux Central, Paris
  - CHU Pontchaillou, Rennes
  - Hôpital Civil, Strasbourg
  - CHU de Toulouse, Hôpital Purpan, Toulouse
- Germany (12):
  - Klinik und Poliklinik für Neurologie, Universitätsklinikum Bonn, Bonn, DE
  - Universitätsklinik Carl Gustav Carus Dresden, Dresden
  - Klinikum der JW Goethe Universität, Frankfurt am Main
  - Asklepios Klinik Barmbek, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Oberhavel Klinicum GmbH - Krankenhaus Hennigsdorf, Hennigsdorf
  - Klinikum Ingolstadt, Ingolstadt
  - Jüdisches Krankenhaus Berlin, Mitte
  - Klinikum rechts der Isar, München
  - Medizinische Fakultät der Universität Rostock,Zentrum für Nervenheilkunde, Rostock
  - Universitätsklinikum Ulm, Klinik für Neurologie im RKU, Ulm
  - Fachkrankenhaus Hubertusburg GmbH, Klinik für Neurologie und Neurologische Intensivmedizin, Wermsdorf
- Israel (3):
  - Hadassah Medical Center Ein Karem, Ein Karem, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Sourasky Tel Aviv Medical Center, Tel Aviv
- Italy (4):
  - Università di Cagliari, Cagliari
  - Ospedale S. Antonio Abate di Gallarate, Gallarate (Varese)
  - Ospedale S. Luigi Gonzaga, Orbassano (TO)
  - Universita Degli Studi di Roma "La Sapienza", Roma
- Mexico (2):
  - Unidad de Investigación en Salud, Chihuahua, CHH
  - Medica Sur, Mexico City, DFE
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Orbis Medisch Concern, Sittard-Geleen
- Poland (5):
  - Centrum Neurologii Klinicznej Sp. Zo.o., Krakow
  - Samodzielny Publiczny ZOZ, Uniwersytecki Szpital Kliniczny Nr1 im. Norberta Barlickiego, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwersytetu Med. im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Institute of Psychiatry and Neurology/Instytut Psychiatrii i Neurologii, Warsaw
- Russia (13):
  - Research Medical Complex "Your Health" Ltd, Kazan'
  - Moscow State Public Medical Institution Clinical Hospital #11, Neurology Department, Moscow
  - Neurology Research Center under the Russian Academy of Medical Sciences, Moscow
  - Russian State Medical University, Department of Neurology and Neurosurgery, Moscow
  - Municipal Treatment and Prevention Institution, City Hospital #33, Nizhny Novgorod
  - Federal State Public Medical Institution: Siberian District Medical Center under the Federal Agency, Novosibirsk
  - Municipal Public Medical Institution: City Hospital #2 of Pyatigorsk, Neurology Department, Pyatigorsk
  - Institute of Human Brain RAS, Laboratory of Neuroimmunology, Saint Petersburg
  - St Petersburg State Pavlov Medical University, Dept of Neurology and Neurosurgery with a Hospital, Saint Petersburg
  - St. Petersburg General Hospital #2, Neurology Department #2, Saint Petersburg
  - St. Petersburg State Public Medical Institution: Nikolayevskaya Hospital, Saint Petersburg
  - Samara Regional Clinical Hospital n.a. Kalinin, Samara
  - State Public Medical Institution: Republican Clinical Hospital n.a. G.G. Kuvatov, Ufa
- Serbia (5):
  - Clinical Centre Serbia, Institute of Neurology,Dr.Subotica 6,Belgrade, Belgrade
  - Military Medical Academy, Institute of Neurology, Belgrade
  - Clinical Centre Kragujevac, Clinic of Neurology, Kragujevac
  - Clinical Centre Nis, Clinic of Neurology, Niš
  - Clinical Centre Vojvodina, Novi Sad
- Spain (4):
  - Hospital Universitario Vall d' Hebron, Barcelona
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Carlos Haya, Neurology Service, Málaga
  - Hospital Virgen Macarena, Seville
- Sweden (2):
  - SU/Östra sjukhuset, Gothenburg
  - Norrlands Universitets sjukhus, Umeå
- Ukraine (4):
  - Institute of Neurology, Psychiatry and Narcology under the AMS of Ukraine, Dep of Neuroinfection& MS, Kharkiv
  - Kiev Municipal Clinical Hospital #4, Department of Demyelinating Diseases of the Nervous System, Kiev
  - Hospital of Directorate of the Medical Corps within the Ukrainian Security Service, Neurology Dept., Kiev-21
  - Lviv National Medical University n.a. Danylo Galytsky, Department of Neurology, Lviv
- United Kingdom (6):
  - Frenchay Hospital, Bristol
  - Addenbrookes Hospital, Cambridge
  - University Hospital of Wales, Dept of Neurology, Cardiff
  - Royal London Hospital, London
  - Salford Royal NHS Foundation Trust, Salford
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Background] CAMMS223 Trial Investigators; Coles AJ, Compston DA, Selmaj KW, Lake SL, Moran S, Margolin DH, Norris K, Tandon PK. Alemtuzumab vs. interferon beta-1a in early multiple sclerosis. N Engl J Med. 2008 Oct 23;359(17):1786-801. doi: 10.1056/NEJMoa0802670. PMID 18946064
- [Background] Cohen JA, Coles AJ, Arnold DL, Confavreux C, Fox EJ, Hartung HP, Havrdova E, Selmaj KW, Weiner HL, Fisher E, Brinar VV, Giovannoni G, Stojanovic M, Ertik BI, Lake SL, Margolin DH, Panzara MA, Compston DA; CARE-MS I investigators. Alemtuzumab versus interferon beta 1a as first-line treatment for patients with relapsing-remitting multiple sclerosis: a randomised controlled phase 3 trial. Lancet. 2012 Nov 24;380(9856):1819-28. doi: 10.1016/S0140-6736(12)61769-3. Epub 2012 Nov 1. PMID 23122652
- [Background] Coles AJ, Twyman CL, Arnold DL, Cohen JA, Confavreux C, Fox EJ, Hartung HP, Havrdova E, Selmaj KW, Weiner HL, Miller T, Fisher E, Sandbrink R, Lake SL, Margolin DH, Oyuela P, Panzara MA, Compston DA; CARE-MS II investigators. Alemtuzumab for patients with relapsing multiple sclerosis after disease-modifying therapy: a randomised controlled phase 3 trial. Lancet. 2012 Nov 24;380(9856):1829-39. doi: 10.1016/S0140-6736(12)61768-1. Epub 2012 Nov 1. PMID 23122650
- [Derived] Ziemssen T, Bass AD, Van Wijmeersch B, Eichau S, Richter S, Hoffmann F, Armstrong NM, Chirieac M, Cunha-Santos J, Singer BA. Long-term efficacy and safety of alemtuzumab in participants with highly active MS: TOPAZ clinical trial and interim analysis of TREAT-MS real-world study. Ther Adv Neurol Disord. 2025 Feb 10;18:17562864241306575. doi: 10.1177/17562864241306575. eCollection 2025. PMID 39935588
- [Derived] Coles AJ, Achiron A, Traboulsee A, Singer BA, Pozzilli C, Oreja-Guevara C, Giovannoni G, Comi G, Freedman MS, Ziemssen T, Shiota D, Rawlings AM, Wong AT, Chirieac M, Montalban X. Safety and efficacy with alemtuzumab over 13 years in relapsing-remitting multiple sclerosis: final results from the open-label TOPAZ study. Ther Adv Neurol Disord. 2023 Sep 21;16:17562864231194823. doi: 10.1177/17562864231194823. eCollection 2023. PMID 37745914
- [Derived] Dayan CM, Lecumberri B, Muller I, Ganesananthan S, Hunter SF, Selmaj KW, Hartung HP, Havrdova EK, LaGanke CC, Ziemssen T, Van Wijmeersch B, Meuth SG, Margolin DH, Poole EM, Baker DP, Senior PA. Endocrine and multiple sclerosis outcomes in patients with autoimmune thyroid events in the alemtuzumab CARE-MS studies. Mult Scler J Exp Transl Clin. 2023 Jan 3;9(1):20552173221142741. doi: 10.1177/20552173221142741. eCollection 2023 Jan-Mar. PMID 36619856
- [Derived] Coles AJ, Jones JL, Vermersch P, Traboulsee A, Bass AD, Boster A, Chan A, Comi G, Fernandez O, Giovannoni G, Kubala Havrdova E, LaGanke C, Montalban X, Oreja-Guevara C, Piehl F, Wiendl H, Ziemssen T. Autoimmunity and long-term safety and efficacy of alemtuzumab for multiple sclerosis: Benefit/risk following review of trial and post-marketing data. Mult Scler. 2022 Apr;28(5):842-846. doi: 10.1177/13524585211061335. Epub 2021 Dec 9. PMID 34882037
- [Derived] Kuhle J, Daizadeh N, Benkert P, Maceski A, Barro C, Michalak Z, Sormani MP, Godin J, Shankara S, Samad TA, Jacobs A, Chung L, Rӧsch N, Kaiser C, Mitchell CP, Leppert D, Havari E, Kappos L. Sustained reduction of serum neurofilament light chain over 7 years by alemtuzumab in early relapsing-remitting MS. Mult Scler. 2022 Apr;28(4):573-582. doi: 10.1177/13524585211032348. Epub 2021 Aug 11. PMID 34378446
- [Derived] Coles AJ, Arnold DL, Bass AD, Boster AL, Compston DAS, Fernandez O, Havrdova EK, Nakamura K, Traboulsee A, Ziemssen T, Jacobs A, Margolin DH, Huang X, Daizadeh N, Chirieac MC, Selmaj KW. Efficacy and safety of alemtuzumab over 6 years: final results of the 4-year CARE-MS extension trial. Ther Adv Neurol Disord. 2021 Apr 23;14:1756286420982134. doi: 10.1177/1756286420982134. eCollection 2021. PMID 34035833
- [Derived] Bass AD, Arroyo R, Boster AL, Boyko AN, Eichau S, Ionete C, Limmroth V, Navas C, Pelletier D, Pozzilli C, Ravenscroft J, Sousa L, Tintore M, Uitdehaag BMJ, Baker DP, Daizadeh N, Choudhry Z, Rog D; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ investigators. Alemtuzumab outcomes by age: Post hoc analysis from the randomized CARE-MS studies over 8 years. Mult Scler Relat Disord. 2021 Apr;49:102717. doi: 10.1016/j.msard.2020.102717. Epub 2020 Dec 24. PMID 33476880
- [Derived] Horakova D, Boster A, Bertolotto A, Freedman MS, Firmino I, Cavalier SJ, Jacobs AK, Thangavelu K, Daizadeh N, Poole EM, Baker DP, Margolin DH, Ziemssen T; CARE-MS I, CARE-MS II, and CAMMS03409 Investigators. Proportion of alemtuzumab-treated patients converting from relapsing-remitting multiple sclerosis to secondary progressive multiple sclerosis over 6 years. Mult Scler J Exp Transl Clin. 2020 Dec 18;6(4):2055217320972137. doi: 10.1177/2055217320972137. eCollection 2020 Oct-Dec. PMID 33414927
- [Derived] Ziemssen T, Bass AD, Berkovich R, Comi G, Eichau S, Hobart J, Hunter SF, LaGanke C, Limmroth V, Pelletier D, Pozzilli C, Schippling S, Sousa L, Traboulsee A, Uitdehaag BMJ, Van Wijmeersch B, Choudhry Z, Daizadeh N, Singer BA; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ investigators. Efficacy and Safety of Alemtuzumab Through 9 Years of Follow-up in Patients with Highly Active Disease: Post Hoc Analysis of CARE-MS I and II Patients in the TOPAZ Extension Study. CNS Drugs. 2020 Sep;34(9):973-988. doi: 10.1007/s40263-020-00749-x. PMID 32710396
- [Derived] Gilmore W, Lund BT, Li P, Levy AM, Kelland EE, Akbari O, Groshen S, Cen SY, Pelletier D, Weiner LP, Javed A, Dunn JE, Traboulsee AL. Repopulation of T, B, and NK cells following alemtuzumab treatment in relapsing-remitting multiple sclerosis. J Neuroinflammation. 2020 Jun 15;17(1):189. doi: 10.1186/s12974-020-01847-9. PMID 32539719
- [Derived] Comi G, Alroughani R, Boster AL, Bass AD, Berkovich R, Fernandez O, Kim HJ, Limmroth V, Lycke J, Macdonell RA, Sharrack B, Singer BA, Vermersch P, Wiendl H, Ziemssen T, Jacobs A, Daizadeh N, Rodriguez CE, Traboulsee A; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ Investigators. Efficacy of alemtuzumab in relapsing-remitting MS patients who received additional courses after the initial two courses: Pooled analysis of the CARE-MS, extension, and TOPAZ studies. Mult Scler. 2020 Dec;26(14):1866-1876. doi: 10.1177/1352458519888610. Epub 2019 Nov 25. PMID 31762387
- [Derived] Van Wijmeersch B, Singer BA, Boster A, Broadley S, Fernandez O, Freedman MS, Izquierdo G, Lycke J, Pozzilli C, Sharrack B, Steingo B, Wiendl H, Wray S, Ziemssen T, Chung L, Margolin DH, Thangavelu K, Vermersch P. Efficacy of alemtuzumab over 6 years in relapsing-remitting multiple sclerosis patients who relapsed between courses 1 and 2: Post hoc analysis of the CARE-MS studies. Mult Scler. 2020 Nov;26(13):1719-1728. doi: 10.1177/1352458519881759. Epub 2019 Nov 1. PMID 31675266
- [Derived] Okai AF, Amezcua L, Berkovich RR, Chinea AR, Edwards KR, Steingo B, Walker A, Jacobs AK, Daizadeh N, Williams MJ; CARE-MS I, CARE-MS II, CAMMS03409, and TOPAZ Investigators. Efficacy and Safety of Alemtuzumab in Patients of African Descent with Relapsing-Remitting Multiple Sclerosis: 8-Year Follow-up of CARE-MS I and II (TOPAZ Study). Neurol Ther. 2019 Dec;8(2):367-381. doi: 10.1007/s40120-019-00159-2. Epub 2019 Oct 25. PMID 31654272
- [Derived] Arroyo R, Bury DP, Guo JD, Margolin DH, Melanson M, Daizadeh N, Cella D. Impact of alemtuzumab on health-related quality of life over 6 years in CARE-MS II trial extension patients with relapsing-remitting multiple sclerosis. Mult Scler. 2020 Jul;26(8):955-963. doi: 10.1177/1352458519849796. Epub 2019 May 30. PMID 31144568
- [Derived] Havrdova E, Arnold DL, Cohen JA, Hartung HP, Fox EJ, Giovannoni G, Schippling S, Selmaj KW, Traboulsee A, Compston DAS, Margolin DH, Thangavelu K, Rodriguez CE, Jody D, Hogan RJ, Xenopoulos P, Panzara MA, Coles AJ; CARE-MS I and CAMMS03409 Investigators. Alemtuzumab CARE-MS I 5-year follow-up: Durable efficacy in the absence of continuous MS therapy. Neurology. 2017 Sep 12;89(11):1107-1116. doi: 10.1212/WNL.0000000000004313. Epub 2017 Aug 23. PMID 28835401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study enrolled participants from previous 3 studies: CAMMS223 (NCT00050778), CAMMS323 (NCT00530348), and CAMMS324 (NCT00548405). Participants were enrolled in this study only after their Month 24 visit in CAMMS323 and CAMMS324. CAMMS223 participants were enrolled within 6 months once their site received approval of extension study.
Pre-assignment Details: Efficacy outcome data was analyzed only on CAMMS323 and CAMMS324 participants; safety data was analyzed on all participants, as pre-specified in protocol.
Groups:
- Alemtuzumab: Participants enrolled from any of the prior studies received long-term follow-up in this study. Participants randomized to receive interferon beta-1a (IFNB-1a) in prior studies received alemtuzumab 12 mg/day infusion intravenously (IV) once daily (QD) for 5 consecutive days in treatment Course 1, and for 3 consecutive days in treatment Course 2, 12 months later in this study. Participants who received 2 treatment courses with alemtuzumab could be treated with additional alemtuzumab courses of 12 mg/day infusion IV QD, for 3 consecutive days at least 48 weeks after the prior course if they had documented evidence of resumed disease activity (defined as >=1 protocol-defined relapse and/or >=2 new or enlarging brain or spinal lesions on magnetic resonance imaging [MRI]), unless they met safety-related retreatment disqualifying criteria.
Period: Overall Study
Arm/Group | Alemtuzumab
Started | 1314
Participants Entered From CAMMS223 | 141
Participants Entered From CAMMS323 | 488
Participants Entered From CAMMS324 | 685
Completed | 1091
Not Completed | 223
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 7
Not completed — Physician Decision | 39
Not completed — Protocol Violation | 1
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 88
Not completed — Lost to Follow-up | 25
Not completed — Death | 9
Not completed — Study terminated by sponsor | 24
Not completed — Other than specified above | 28

BASELINE CHARACTERISTICS:
Groups:
- Alemtuzumab: Participants enrolled from any of the previous studies received long-term follow-up in this study. Participants randomized to receive IFNB-1a in any of the previous studies received alemtuzumab 12 mg/day infusion IV, QD for 5 consecutive days in treatment Course 1, and for 3 consecutive days in treatment Course 2, 12 months later in this study. Participants who received 2 treatment courses with alemtuzumab could be treated with additional alemtuzumab courses of 12 mg/day infusion IV QD, for 3 consecutive days at least 48 weeks after the prior course if they had documented evidence of resumed disease activity (defined as >=1 protocol-defined relapse and/or >=2 new or enlarging brain or spinal lesions on MRI), unless they met safety-related retreatment disqualifying criteria.
Arm/Group | Alemtuzumab
Number analyzed (Participants) | 1314
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 857
  Male | 457

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR)
Description: Relapse was defined as new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination, attributable to multiple sclerosis (MS) that last for at least 48 hours, present at normal body temperature, and that were preceded by at least 30 days of clinical stability. ARR was obtained from the total number of confirmed relapses that occurred during the treatment follow-up time of all participants divided by the sum of follow-up time of all participants involved in certain treatment groups. ARR was estimated through negative binomial regression with robust variance estimation.
Time Frame: Year 3, 4, 5, 6 from the Baseline (Month 0 of CAMMS323 and Month 0 of CAMMS324 for "Alemtuzumab Treatment CAMMS323 Extension" group and "Alemtuzumab Treatment CAMMS324 Extension" group, respectively)
Population: Subset of full analysis set (FAS - defined as all participants randomized in CAMMS223, CAMMS323, and CAMMS324 and who received at least 1 dose of study drug) included participants who had received at least 1 dose of alemtuzumab in CAMMS323 and CAMMS324. Number of participants analyzed = participants with available data for this outcome measure.
Measure: Number; unit: relapses per participant per year
Groups:
- Alemtuzumab Treatment CAMMS323 Extension: Participants who were randomized to alemtuzumab 12 mg/day treatment in CAMMS323 (NCT00530348) and enrolled in this extension study (CAMMS03409).
- Alemtuzumab Treatment CAMMS324 Extension: Participants who were randomized to alemtuzumab 12 mg/day treatment in CAMMS324 (NCT00548405) and enrolled in this extension study (CAMMS03409).
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 353 | 391
relapses per participant per year
  Year 3 | 0.19 | 0.22
  Year 4 | 0.16 | 0.24
  Year 5 | 0.15 | 0.19
  Year 6 | 0.12 | 0.16

2. Primary Outcome: Annualized Relapse Rate (ARR) Before and After Receiving Alemtuzumab
Description: Relapse was defined as new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination, attributable to MS that last for at least 48 hours, present at normal body temperature, and that were preceded by at least 30 days of clinical stability. ARR was obtained from the total number of confirmed relapses that occurred during the treatment follow-up time of all participants divided by the sum of total follow-up time of all participants involved in certain treatment groups. ARR was estimated through repeated negative binomial regression with robust variance estimation and covariate adjustment for geographic region. The IFNB-1a/Alemtuzumab switch from CAMMS323 or CAMMS324 to CAMMS03409 pre alemtuzumab reporting group consisted of the same participants as those in the corresponding post alemtuzumab reporting group.
Time Frame: Baseline (Year 0 of initial studies) up to Year 4
Population: Subset of FAS who received IFNB-1a in CAMMS323 or CAMMS324 and who were treated with alemtuzumab in CAMMS03409.
Measure: Number (95% Confidence Interval); unit: relapses per participant per year
Groups:
- IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab): Participants who received IFNB-1a in CAMMS323, were treated with alemtuzumab in CAMMS03409. IFNB-1a treatment period
- IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab): Participants who received IFNB-1a in CAMMS323, were treated with alemtuzumab in CAMMS03409. Alemtuzumab treatment period
- IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab): Participants who received IFNB-1a in CAMMS324, were treated with alemtuzumab in CAMMS03409. IFNB-1a treatment period
- IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab): Participants who received IFNB-1a in CAMMS324, were treated with alemtuzumab in CAMMS03409. Alemtuzumab treatment period
Arm/Group | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab)
Number analyzed (Participants) | 139 | 139 | 143 | 143
relapses per participant per year | 0.42 [0.28 to 0.64] | 0.14 [0.09 to 0.21] | 0.60 [0.45 to 0.78] | 0.15 [0.10 to 0.22]

3. Primary Outcome: Annualized Relapse Rate (ARR) Before and After Alemtuzumab Retreatment
Description: Relapse was defined as new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination, attributable to MS that last for at least 48 hours, present at normal body temperature, and that were preceded by at least 30 days of clinical stability. ARR was obtained from the total number of confirmed relapses that occurred during the treatment follow-up time of all participants divided by the sum of total follow-up time of all participants involved in certain treatment groups. ARR was estimated through negative binomial regression with robust variance estimation without covariate adjustment.
Time Frame: Year 1 prior to retreatment, Year 1, 2, 3 after retreatment
Population: Subset of FAS included participants who had received alemtuzumab in CAMMS323 or CAMMS324 and received an additional course of alemtuzumab in this extension study.
Measure: Number (95% Confidence Interval); unit: relapses per participant per year
Groups:
- Alemtuzumab Retreatment: Participants who received alemtuzumab in CAMMS323 (NCT00530348) or CAMMS324 (NCT00548405), received an additional course of alemtuzumab in this study.
Arm/Group | Alemtuzumab Retreatment
Number analyzed (Participants) | 321
relapses per participant per year
  Year 1 prior to retreatment | 0.79 [0.73 to 0.87]
  Year 1 after retreatment | 0.18 [0.14 to 0.24]
  Year 2 after retreatment | 0.29 [0.23 to 0.38]
  Year 3 after retreatment | 0.30 [0.21 to 0.41]

4. Primary Outcome: Number of Participants With Sustained Accumulation of Disability (SAD)
Description: SAD: defined as an increase of at least 1.5 points in Expanded Disability Status Scale (EDSS) score for participants with prior study baseline score of 0 and increase of at least 1.0 point for participants with a prior study baseline score of 1.0 or more; and the increase persisted over a 6-month consecutive period. EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) and ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), higher scores indicating worse neurological function. Number of participants with SAD was estimated by Kaplan-Meier method and reported in this outcome measure. Baseline was defined as Year 0 of CAMMS323 and Year 0 of CAMMS324 for "alemtuzumab treatment CAMMS323 extension" group and "alemtuzumab Treatment CAMMS324 Extension" group, respectively.
Time Frame: Baseline (Year 0) up to Year 6
Population: Subset of full analysis set (FAS - defined as all participants randomized in CAMMS223, CAMMS323, and CAMMS324 and who received at least 1 dose of study drug) included participants who had received at least 1 dose of alemtuzumab in CAMMS323 and CAMMS324.
Measure: Count of Participants; unit: Participants
Groups:
- Alemtuzumab Treatment CAMMS323 Extension: Participants who were randomized to alemtuzumab 12 mg/day treatment in CAMMS323 (NCT00530348) and enrolled in this extension study.
- Alemtuzumab Treatment CAMMS324 Extension: Participants who were randomized to alemtuzumab 12 mg/day treatment in CAMMS324 (NCT00548405) and enrolled in this extension study.
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 376 | 426
Participants | 79 | 118
Statistical Analysis 1: Comparison: Alemtuzumab Treatment CAMMS323 Extension; Test type: Superiority or Other; Percentage with SAD = 22.33, 95% CI 2-sided [18.33 to 27.06] — The percentage and 95% CI of the participants with SAD are estimated by the Kaplan Meier method
Statistical Analysis 2: Comparison: Alemtuzumab Treatment CAMMS324 Extension; Test type: Superiority or Other; Percentage with SAD = 29.69, 95% CI 2-sided [25.42 to 34.49] — The percentage and 95% CI of the participants with SAD are estimated by the Kaplan Meier method

5. Primary Outcome: Number of Participants With Sustained Accumulation of Disability (SAD) Before and After Alemtuzumab Treatment: 2 Year Comparison
Description: SAD: defined as an increase of at least 1.5 points in EDSS score for participants with prior study baseline score of 0 and increase of at least 1.0 point for participants with a prior study baseline score of 1.0 or more; and the increase persisted over a 6-month consecutive period. EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) and ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), higher scores indicating worse neurological function. Number of participants with SAD over 2 years before and 2 years after alemtuzumab treatment were estimated by Kaplan-Meier method and reported in this outcome measure. The IFNB-1a/Alemtuzumab switch pre alemtuzumab reporting group consisted of the same participants as those in the corresponding post alemtuzumab reporting group.
Time Frame: Baseline (Year 0 of initial studies) up to Year 4
Population: Subset of FAS who received IFNB-1a in CAMMS323 or CAMMS324 and who were treated with alemtuzumab in CAMMS03409.
Measure: Count of Participants; unit: Participants
Groups:
- IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab): Participants who received IFNB-1a in CAMMS323 who were treated with alemtuzumab in CAMMS03409. IFNB-1a treatment period
- IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab): Participants who received IFNB-1a in CAMMS323 who were treated with alemtuzumab in CAMMS03409. Alemtuzumab treatment period
- IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab): Participants who received IFNB-1a in CAMMS324 who were treated with alemtuzumab in CAMMS03409. IFNB-1a treatment period
- IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab): Participants who received IFNB-1a in CAMMS324 who were treated with alemtuzumab in CAMMS03409. Alemtuzumab treatment period
Arm/Group | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab)
Number analyzed (Participants) | 139 | 139 | 143 | 143
Participants | 13 | 11 | 29 | 17
Statistical Analysis 1: Comparison: IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab); Test type: Superiority or Other; Percentage with SAD = 9.35, 95% CI 2-sided [5.54 to 15.56] — The percentage and 95% CI of the participants with SAD are estimated by the Kaplan Meier method
Statistical Analysis 2: Comparison: IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab); Test type: Superiority or Other; Percentage with SAD = 7.95, 95% CI 2-sided [4.48 to 13.90] — The percentage and 95% CI of the participants with SAD are estimated by the Kaplan Meier method
Statistical Analysis 3: Comparison: IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab); Test type: Superiority or Other; Percentage with SAD = 20.42, 95% CI 2-sided [14.67 to 28.03] — The percentage and 95% CI of the participants with SAD are estimated by the Kaplan Meier method
Statistical Analysis 4: Comparison: IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab); Test type: Superiority or Other; Percentage with SAD = 11.99, 95% CI 2-sided [7.63 to 18.58] — The percentage and 95% CI of the participants with SAD are estimated by the Kaplan Meier method

6. Secondary Outcome: Number of Participants With Sustained Reduction in Disability (SRD) Assessed by EDSS at Year 6
Description: SRD was defined as a ≥1 point decrease in EDSS score lasting >= 6 months. SRD is only applicable to participants with a baseline EDSS score of >= 2.0. EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicate worse neurological function. Number of participants with SRD at Year 6 was estimated using Kaplan-Meier method and reported in this outcome measure.
Time Frame: Baseline (Year 0) up to Year 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 235 | 321
Participants | 74 | 130
Statistical Analysis 1: Comparison: Alemtuzumab Treatment CAMMS323 Extension; Test type: Superiority or Other; Percentage with SRD = 32.69, 95% CI 2-sided [26.96 to 39.28] — The percentage and 95% CI of the participants with SRD are estimated by the Kaplan Meier method
Statistical Analysis 2: Comparison: Alemtuzumab Treatment CAMMS324 Extension; Test type: Superiority or Other; Percentage with SRD = 42.46, 95% CI 2-sided [37.08 to 48.28] — The percentage and 95% CI of the participants with SRD are estimated by the Kaplan Meier method

7. Secondary Outcome: Number of Participants With Sustained Reduction in Disability (SRD) Assessed by EDSS (After Alemtuzumab Treatment) at Year 2 of the Extension Study
Description: SRD was defined as a >=1 point decrease in EDSS score lasting >=6 months. SRD is only applicable to participants with a baseline EDSS score of ≥2.0. EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicate worse neurological function. Number of participants with SRD at Year 2 of CAMMS03409 was estimated using Kaplan-Meier method and reported in this outcome measure. The IFNB-1a/Alemtuzumab switch from CAMMS323 or CAMMS324 to CAMMS03409 pre alemtuzumab reporting group consisted of the same participants as those in the corresponding post alemtuzumab reporting group.
Time Frame: Extension study (CAMMS03409) baseline up to Extension Year 2
Population: Subset of FAS who received IFNB-1a in CAMMS323 or CAMMS324 and who were treated with alemtuzumab in CAMMS03409. Number of participants analyzed = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab)
Number analyzed (Participants) | 65 | 102
Participants | 11 | 14
Statistical Analysis 1: Comparison: IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab); Test type: Superiority or Other; Percentage with SRD = 16.92, 95% CI 2-sided [9.75 to 28.47] — The percentage and 95% CI of the participants with SRD are estimated by the Kaplan Meier method
Statistical Analysis 2: Comparison: IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab); Test type: Superiority or Other; Percentage with SRD = 13.89, 95% CI 2-sided [8.47 to 22.33] — The percentage and 95% CI of the participants with SRD are estimated by the Kaplan Meier method

8. Secondary Outcome: Change From Initial Study Baseline in EDSS Score at Year 3, 4, 5 and 6
Description: EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicate worse neurological function. Change was calculated by subtracting baseline (Month 0 of the study CAMMS323 [NCT00530348] or CAMMS324 [NCT00548405]) value from EDSS scores at specified time points.
Time Frame: Baseline (Month 0 of CAMMS323 and Month 0 of CAMMS324 for "Alemtuzumab Treatment CAMMS323 Extension" group and "Alemtuzumab Treatment CAMMS324 Extension" group, respectively), Year 3, 4, 5, 6
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Alemtuzumab Treatment CAMMS323 Extension: Participants who were randomized to alemtuzumab 12 mg/day treatment in CAMMS323 (NCT00530348) and enrolled in extension study CAMMS03409.
- Alemtuzumab Treatment CAMMS324 Extension: Participants who were randomized to alemtuzumab 12 mg/day treatment in CAMMS324 (NCT00548405) and enrolled in extension study CAMMS03409.
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 326 | 370
units on a scale
  Change at Year 3 | -0.08 [-0.20 to 0.04] | -0.02 [-0.14 to 0.10]
  Change at Year 4 | -0.06 [-0.19 to 0.07] | 0.06 [-0.07 to 0.19]
  Change at Year 5 | 0.06 [-0.08 to 0.19] | 0.13 [-0.01 to 0.27]
  Change at Year 6 | 0.09 [-0.04 to 0.23] | 0.18 [0.03 to 0.32]

9. Secondary Outcome: Change From Initial Study Baseline in EDSS Score Before and After Alemtuzumab Treatment: 2 Year Comparison
Description: EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicate worse neurological function. Change was calculated by subtracting baseline (Month 0 of the study CAMMS323 or CAMMS324 for pre alemtuzumab period or CAMMS03409 baseline for post alemtuzumab period) value, from EDSS scores at specified time points. The IFNB-1a/Alemtuzumab switch pre alemtuzumab reporting group consisted of the same participants as those in the corresponding post alemtuzumab reporting groups. Baseline was defined as Year 0 of CAMMS323 and Year 0 of CAMMS324 for "CAMMS323 participants" and "CAMMS324 participants" respectively.
Time Frame: Baseline (Year 0 of initial studies) up to Year 4
Population: Subset of FAS who received IFNB-1a in CAMMS323 or CAMMS324 and who were treated with alemtuzumab in CAMMS03409.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab)
Number analyzed (Participants) | 139 | 139 | 143 | 143
units on a scale
  Year 0 - 2 | -0.15 [-0.32 to 0.03] | -0.07 [-0.23 to 0.09] | 0.11 [-0.05 to 0.26] | -0.02 [-0.18 to 0.14]
  Year 3 - 4 | -0.21 [-0.43 to 0.00] | 0.08 [-0.11 to 0.27] | 0.20 [-0.01 to 0.41] | 0.13 [-0.05 to 0.31]

10. Secondary Outcome: Change From Retreatment Baseline in EDSS Score After Alemtuzumab Retreatment
Description: EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS), where higher scores indicate worse neurological function. Change was calculated by subtracting retreatment baseline (annual visit prior to the retreatment start date) value from EDSS scores at specified time points.
Time Frame: Retreatment baseline, Year 1, 2 and 3 after retreatment baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Alemtuzumab Retreatment: Participants who received alemtuzumab in CAMMS323 or CAMMS324 who received an additional course of alemtuzumab in CAMMS03409.
Arm/Group | Alemtuzumab Retreatment
Number analyzed (Participants) | 321
units on a scale
  Retreatment baseline: number analyzed (Participants) | 307
  Retreatment baseline | 2.89 (1.514)
  Change at Year 1 after retreatment baseline: number analyzed (Participants) | 256
  Change at Year 1 after retreatment baseline | -0.22 (1.033)
  Change at Year 2 after retreatment baseline: number analyzed (Participants) | 158
  Change at Year 2 after retreatment baseline | -0.13 (1.109)
  Change at Year 3 after retreatment baseline: number analyzed (Participants) | 75
  Change at Year 3 after retreatment baseline | 0.07 (1.356)

11. Secondary Outcome: Percentage of Participants Without New or Enlarging Magnetic Resonance Imaging (MRI)-T2-Hypertense Lesion Activity
Description: Analysis of new or enlarging lesions that appear hyperintense on T2-weighted MRI scans performed annually.
Time Frame: Year 3, 4, 5 and 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 328 | 356
percentage of participants
  Year 3 | 72.6 | 68.8
  Year 4: number analyzed (Participants) | 323 | 332
  Year 4 | 70.3 | 70.2
  Year 5: number analyzed (Participants) | 319 | 321
  Year 5 | 70.2 | 67.0
  Year 6: number analyzed (Participants) | 307 | 312
  Year 6 | 66.8 | 69.6

12. Secondary Outcome: Percentage of Participants Without New or Enlarging MRI-T2-Hypertense Lesion Activity Before and After Alemtuzumab Treatment
Description: Analysis of new or enlarging lesions that appear hyperintense on T2-weighted MRI scans performed annually. The IFNB-1a/Alemtuzumab switch from CAMMS323 or CAMMS324 to CAMMS03409 pre alemtuzumab reporting group consisted of the same participants as those in the corresponding post alemtuzumab reporting group.
Time Frame: Baseline (Year 0 of initial studies) up to Year 4
Population: Subset of FAS who received IFNB-1a in CAMMS323 or CAMMS324 and who were treated with alemtuzumab in CAMMS03409.
Measure: Number; unit: percentage of participants
Arm/Group | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab)
Number analyzed (Participants) | 139 | 139 | 143 | 143
percentage of participants
  Year 0 - 1: number analyzed (Participants) | 135 | 135 | 139 | 138
  Year 0 - 1 | 57 | 79.3 | 44.6 | 63.8
  Year 0 - 2: number analyzed (Participants) | 135 | 132 | 139 | 131
  Year 0 - 2 | 60.7 | 81.8 | 47.5 | 81.7

13. Secondary Outcome: Percentage of Participants Without New or Enlarging MRI-T2-Hypertense Lesion Activity Before and After Alemtuzumab Retreatment
Description: Analysis of new or enlarging lesions that appear hyperintense on T2-weighted MRI scans performed annually. Retreatment baseline was the annual visit prior to the retreatment start date.
Time Frame: Retreatment Baseline, Year 1, 2 and 3 after retreatment
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Alemtuzumab Retreatment
Number analyzed (Participants) | 321
percentage of participants
  Retreatment baseline: number analyzed (Participants) | 315
  Retreatment baseline | 49.2
  Year 1 after retreatment baseline: number analyzed (Participants) | 301
  Year 1 after retreatment baseline | 64.1
  Year 2 after retreatment baseline: number analyzed (Participants) | 197
  Year 2 after retreatment baseline | 66.0
  Year 3 after retreatment baseline: number analyzed (Participants) | 113
  Year 3 after retreatment baseline | 60.2

14. Secondary Outcome: Percentage Change From Baseline in MRI-T2-Hypertense Lesion Volumes at Year 3, 4, 5, 6
Description: Lesion volume was quantitatively assessed by hyperintensity on T2-weighted MRI scans.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 332 | 364
percent change
  Change at Year 3 | -6.57 (29.96) | 1.69 (31.62)
  Change at Year 4: number analyzed (Participants) | 327 | 339
  Change at Year 4 | -5.04 (32.88) | 4.97 (41.11)
  Change at Year 5: number analyzed (Participants) | 324 | 336
  Change at Year 5 | -4.09 (36.99) | 12.37 (80.74)
  Change at Year 6: number analyzed (Participants) | 309 | 319
  Change at Year 6 | -2.68 (42.92) | 11.46 (73.91)

15. Secondary Outcome: Percentage of Participants Without New Gadolinium-enhancing MRI Lesion Activity
Description: Analysis of new gadolinium-enhancing lesions that appear on MRI scans performed annually. Baseline was the prior annual visit.
Time Frame: Year 3, 4, 5 and 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 330 | 356
percentage of participants
  Year 3 | 90.6 | 86.5
  Year 4: number analyzed (Participants) | 325 | 331
  Year 4 | 87.1 | 88.8
  Year 5: number analyzed (Participants) | 321 | 321
  Year 5 | 87.5 | 89.4
  Year 6: number analyzed (Participants) | 308 | 310
  Year 6 | 86.7 | 90.0

16. Secondary Outcome: Percent Change From Baseline in Brain Parenchymal Fractions (BPF) at Year 3, 4, 5 and 6
Description: Brain parenchymal fraction (calculated as the ratio of brain parenchymal volume to total intradural volume), is a sensitive indicator of brain atrophy.
Time Frame: Baseline (Month 0 of CAMMS323 and Month 0 of CAMMS324 for "Alemtuzumab Treatment CAMMS323 Extension" group and "Alemtuzumab Treatment CAMMS324 Extension" group, respectively), Year 3, 4, 5 and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 325 | 355
percent change
  Change at Year 3 | -1.068 (1.185) | -0.761 (1.240)
  Change at Year 4: number analyzed (Participants) | 323 | 331
  Change at Year 4 | -1.251 (1.228) | -0.949 (1.341)
  Change at Year 5: number analyzed (Participants) | 321 | 317
  Change at Year 5 | -1.437 (1.317) | -0.983 (1.374)
  Change at Year 6: number analyzed (Participants) | 308 | 315
  Change at Year 6 | -1.601 (1.370) | -1.051 (1.472)

17. Secondary Outcome: Percentage of Relapse Free Participants
Description: Relapse was defined as new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination, attributable to MS that last for at least 48 hours, present at normal body temperature, and that were preceded by at least 30 days of clinical stability.
Time Frame: Year 3, 4, 5 and 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 353 | 391
percentage of participants
  Year 3 | 84.14 | 80.56
  Year 4 | 86.84 | 79.27
  Year 5 | 87.35 | 83.29
  Year 6 | 88.96 | 86.86

18. Secondary Outcome: Change From Baseline in Physical Component Score (PCS) of Short Form-36 (SF-36) Health Survey at Year 3, 4, 5 and 6
Description: SF-36 is a participant reported standardized survey designed to assess generic health related quality of life. It consisted of 36 items evaluating 8 aspects of functional health and well-being: 1) physical functioning, 2) role physical, 3) bodily pain, 4) general health, 5) vitality, 6) social functioning, 7) role emotional and 8) mental health. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Scores of first four health aspects (1 - 4) were aggregated to derive the PCS ranging from 0 (worst) to 100 (best), where higher scores indicated good health condition.
Time Frame: Baseline (Month 0 of CAMMS323 and Month 0 of CAMMS324 for "alemtuzumab treatment CAMMS323 extension group", "alemtuzumab Treatment CAMMS324 Extension" group, respectively),Year 3, 4, 5 and 6
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 340 | 375
units on a scale
  Change at Year 3 | 1.90 [0.85 to 2.95] | 1.72 [0.84 to 2.60]
  Change at Year 4 | 2.15 [1.10 to 3.20] | 1.34 [0.40 to 2.28]
  Change at Year 5 | 1.85 [0.75 to 2.94] | 1.34 [0.39 to 2.29]
  Change at Year 6 | 1.65 [0.56 to 2.74] | 1.00 [-0.03 to 2.03]

19. Secondary Outcome: Change From Baseline in Physical Component Score (PCS) of Short Form-36 (SF-36) Health Survey Before and After Alemtuzumab Treatment: 2 Year Comparison
Description: SF-36 is a participant reported standardized survey designed to assess generic health related quality of life. It consisted of 36 items evaluating 8 aspects of functional health and well-being: 1) physical functioning, 2) role physical, 3) bodily pain, 4) general health, 5) vitality, 6) social functioning, 7) role emotional and 8) mental health. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Scores of first four health aspects (1 - 4) were aggregated to derive the PCS ranging from 0 (worst) to 100 (best), where higher scores indicated good health condition. The IFNB-1a/Alemtuzumab switch from CAMMS323 or CAMMS324 to CAMMS03409 pre alemtuzumab reporting group consisted of the same participants as those in the corresponding post alemtuzumab reporting group. Baseline was defined as Year 0 of CAMMS323 and Year 0 of CAMMS324 for "CAMMS323" and "CAMMS324" participants, respectively.
Time Frame: Baseline (Year 0 of initial studies) up to Year 4
Population: Subset of FAS who received IFNB-1a in CAMMS323 or CAMMS324 and who were treated with alemtuzumab in CAMMS03409.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab)
Number analyzed (Participants) | 139 | 139 | 143 | 143
units on a scale
  Year 1 | 1.16 [-0.48 to 2.81] | 2.00 [0.43 to 3.57] | 0.79 [-0.34 to 1.93] | 1.56 [0.38 to 2.75]
  Year 2 | 1.20 [-0.54 to 2.95] | 0.41 [-1.21 to 2.04] | 0.45 [-0.86 to 1.76] | 1.31 [0.14 to 2.48]

20. Secondary Outcome: Change From Baseline in Mental Component Score (MCS) of Short Form-36 (SF-36) at Year 3, 4, 5, and 6
Description: SF-36 is a participant reported standardized survey designed to assess generic health related quality of life. It consisted of 36 items evaluating 8 aspects of functional health and well-being: 1) physical functioning, 2) role physical, 3) bodily pain, 4) general health, 5) vitality, 6) social functioning, 7) role emotional and 8) mental health. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Scores of last four health aspects (5 - 8) were aggregated to derive the MCS ranging from 0 (worst) to 100 (best), where higher scores indicated good health condition.
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 340 | 375
units on a scale
  Change at Year 3 | 2.43 [1.07 to 3.78] | 1.96 [0.85 to 3.07]
  Change at Year 4 | 3.17 [1.85 to 4.49] | 1.91 [0.77 to 3.05]
  Change at Year 5 | 2.54 [1.23 to 3.85] | 1.75 [0.59 to 2.92]
  Change at Year 6 | 2.41 [1.01 to 3.80] | 1.58 [0.35 to 2.82]

21. Secondary Outcome: Change From Baseline in Mental Component Score (MCS) of Short Form-36 (SF-36) Before and After Alemtuzumab Treatment: 2 Year Comparison
Description: SF-36 is a participant reported standardized survey designed to assess generic health related quality of life. It consisted of 36 items evaluating 8 aspects of functional health and well-being: 1) physical functioning, 2) role physical, 3) bodily pain, 4) general health, 5) vitality, 6) social functioning, 7) role emotional and 8) mental health. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Scores of last four health aspects (5 - 8) were aggregated to derive the MCS ranging from 0 (worst) to 100 (best), where higher scores indicated good health condition. The IFNB-1a/Alemtuzumab switch from CAMMS323 or CAMMS324 to CAMMS03409 pre alemtuzumab reporting group consisted of the same participants as those in the corresponding post alemtuzumab reporting group. Baseline was defined as Year 0 of CAMMS323 and Year 0 of CAMMS324 for "CAMMS323" and "CAMMS324" participants, respectively.
Time Frame: Baseline (Year 0 of initial studies) up to Year 4
Population: Subset of FAS who received IFNB-1a in CAMMS323 or CAMMS324 and who were treated with alemtuzumab in CAMMS03409.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab)
Number analyzed (Participants) | 139 | 139 | 143 | 143
units on a scale
  Change at Year 1 | 2.88 [0.49 to 5.27] | 1.98 [-0.46 to 4.43] | 1.83 [0.30 to 3.36] | 1.21 [-0.31 to 2.74]
  Change at Year 2 | 2.32 [-0.11 to 4.74] | 2.08 [-0.38 to 4.54] | 1.65 [0.05 to 3.25] | 1.65 [-0.01 to 3.31]

22. Secondary Outcome: Change From Baseline in Self-reported Quality of Life as Assessed by Functional Assessment of Multiple Sclerosis (FAMS) Score at Year 3, 4, 5 and 6
Description: FAMS is a widely accepted, MS-specific, quality of life questionnaire. It comprised of 58 items on 7 subscales: mobility (7 items); symptoms (7 items); emotional well-being (7 items); general contentment (7 items); thinking and fatigue (9 items); family/social well-being (7 items); and additional concerns (14 items, these are not scored). Participants provided their response based on the recall of past week. Each item was rated on a 5-point scale ranges from 0 (poor) to 4 (best), where higher scores indicated higher/better quality of life. Scores from 44 calculable items were summed to provide FAMS total score. FAMS total score ranges from 0 (poor) to 176 (best), where higher scores indicated higher/better quality of life.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 340 | 372
units on a scale
  Change at Year 3 | 5.28 [2.03 to 8.52] | 4.55 [1.89 to 7.21]
  Change at Year 4 | 6.81 [3.55 to 10.08] | 3.65 [0.98 to 6.32]
  Change at Year 5 | 4.82 [1.55 to 8.10] | 3.57 [0.78 to 6.37]
  Change at Year 6 | 4.40 [1.03 to 7.78] | 3.16 [0.07 to 6.25]

23. Secondary Outcome: Change From Baseline in Self-reported Quality of Life as Assessed by Functional Assessment of Multiple Sclerosis (FAMS) Score Before and After Alemtuzumab Treatment: 2 Year Comparison
Description: FAMS is a widely accepted, MS-specific, quality of life questionnaire. It comprised of 58 items on 7 subscales: mobility (7 items); symptoms (7 items); emotional well-being (7 items); general contentment (7 items); thinking and fatigue (9 items); family/social well-being (7 items); and additional concerns (14 items, these are not scored). Participants provided their response based on the recall of past week. Each item was rated on a 5-point scale ranges from 0 (poor) to 4 (best), where higher scores indicated higher/better quality of life. Scores from 44 calculable items were summed to provide FAMS total score. FAMS total score ranges from 0 (poor) to 176 (best), where higher scores indicated higher/better quality of life. The IFNB-1a/Alemtuzumab switch from CAMMS323 or CAMMS324 to CAMMS03409 pre alemtuzumab reporting group consisted of the same participants as those in the corresponding post alemtuzumab reporting group.
Time Frame: Baseline (Year 0 of initial studies) up to Year 4
Population: Subset of FAS who received IFNB-1a in CAMMS323 or CAMMS324 and who were treated with alemtuzumab in CAMMS03409.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab: Participants who received IFNB-1a in CAMMS323 who were treated with alemtuzumab in CAMMS03409. IFNB-1a treatment period
Arm/Group | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab)
Number analyzed (Participants) | 139 | 139 | 143 | 143
units on a scale
  Change at Year 1 | 4.27 [-1.17 to 9.72] | 4.82 [0.10 to 9.53] | 3.19 [-0.12 to 6.51] | 5.83 [2.74 to 8.92]
  Change at Year 2 | 1.88 [-3.63 to 7.38] | 3.10 [-2.16 to 8.35] | 0.93 [-2.86 to 4.71] | 4.66 [1.07 to 8.24]

24. Secondary Outcome: Change From Baseline in European Quality of Life -5 Dimension (EQ-5D) Visual Analog Scale Score at Year 3, 4, 5 and 6
Description: EQ-5D is a standardized instrument for measuring health status consisting of EQ-5D descriptive system and Visual Analogue Scale (VAS). The EQ-5D VAS range is from 0-100, higher scores indicate a better health state and a positive change indicates improvement.
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Alemtuzumab Treatment CAMMS323 Extension | Alemtuzumab Treatment CAMMS324 Extension
Number analyzed (Participants) | 337 | 374
units on a scale
  Change at Year 3 | 3.505 [1.438 to 5.572] | 2.859 [1.008 to 4.710]
  Change at Year 4 | 5.144 [3.078 to 7.210] | 2.992 [1.145 to 4.838]
  Change at Year 5 | 4.409 [2.303 to 6.515] | 3.034 [1.169 to 4.898]
  Change at Year 6 | 4.134 [1.946 to 6.323] | 3.155 [0.933 to 5.377]

25. Secondary Outcome: Change From Baseline in European Quality of Life -5 Dimension (EQ-5D) Visual Analog Scale Score Before and After Alemtuzumab Treatment: 2 Year Comparison
Description: EQ-5D is a standardized instrument for measuring health status consisting of EQ-5D descriptive system and VAS. The EQ-5D VAS range is from 0-100, higher scores indicate a better health state and a positive change indicates improvement. The IFNB-1a/Alemtuzumab switch from CAMMS323 or CAMMS324 to CAMMS03409 pre alemtuzumab reporting group consisted of the same participants as those in the corresponding post alemtuzumab reporting group.
Time Frame: Baseline (Year 0 of initial studies) up to Year 4
Population: Subset of FAS who received IFNB-1a in CAMMS323 or CAMMS324 and who were treated with alemtuzumab in CAMMS03409.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS323/03409 (Post Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Pre Alemtuzumab) | IFNB-1a/Alemtuzumab Switch CAMMS324/03409 (Post Alemtuzumab)
Number analyzed (Participants) | 139 | 139 | 143 | 143
units on a scale
  Change at Year 1 | 4.165 [0.639 to 7.691] | 4.576 [1.419 to 7.733] | 1.663 [-0.893 to 4.219] | 4.337 [1.614 to 7.059]
  Change at Year 2 | 2.359 [-1.319 to 6.037] | 4.515 [1.407 to 7.622] | -0.712 [-3.552 to 2.129] | 3.346 [0.324 to 6.368]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form in the extension study up to the end of extension study visit (up to Year 6) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events (TEAEs), AEs that developed/worsened during or at any time after first alemtuzumab treatment. Alemtuzumab TEAEs were defined as AEs with start dates and start times on or after the date and time of the first alemtuzumab treatment in CAMMS03409 or in prior studies (CAMMS223, CAMMS323, or CAMMS324).
Groups:
- Alemtuzumab: Participants enrolled in any of the previous studies who had received alemtuzumab. Participants enrolled in any of the previous studies who had received IFNB-1a, who received alemtuzumab 12 mg/day infusion in this study.
Arm/Group | Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 376/1314
Other Adverse Events (participants affected / at risk) | 1225/1314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab (N=1314)
Acquired haemophilia (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Autoimmune pancytopenia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 16
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 3
Angina pectoris (Cardiac disorders) | 4
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 2
Bradycardia foetal (Cardiac disorders) | 1
Bradycardia neonatal (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Congestive cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Pericarditis (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 3
Foetal cystic hygroma (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Autoimmune hypothyroidism (Endocrine disorders) | 1
Autoimmune thyroiditis (Endocrine disorders) | 4
Basedow's disease (Endocrine disorders) | 39
Goitre (Endocrine disorders) | 3
Hyperparathyroidism (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 14
Hypothyroidism (Endocrine disorders) | 4
Cataract (Eye disorders) | 1
Endocrine ophthalmopathy (Eye disorders) | 4
Glaucoma (Eye disorders) | 1
Iridocyclitis (Eye disorders) | 1
Optic atrophy (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Colitis ischaemic (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Duodenitis (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatic fistula (Gastrointestinal disorders) | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Catheter site pain (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Death (General disorders) | 1
Device dislocation (General disorders) | 1
Fatigue (General disorders) | 1
Inflammation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Perforated ulcer (General disorders) | 1
Pyrexia (General disorders) | 2
Biliary dyskinesia (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 4
Cholecystitis acute (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 4
Hepatitis acute (Hepatobiliary disorders) | 1
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 1
Anaphylactoid reaction (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 3
Abscess bacterial (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Appendicitis perforated (Infections and infestations) | 1
Bone abscess (Infections and infestations) | 1
Breast abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 6
Chronic hepatitis C (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 2
Endometritis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 7
Gastroenteritis bacterial (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 2
HIV infection (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 10
Infection (Infections and infestations) | 1
Infectious colitis (Infections and infestations) | 1
Infective myositis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Lung abscess (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pancreas infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 13
Pneumonia fungal (Infections and infestations) | 1
Pneumonia legionella (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 4
Pyelonephritis acute (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 2
Scrotal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 8
Soft tissue infection (Infections and infestations) | 1
Staphylococcal abscess (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Tubo-ovarian abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 7
Urosepsis (Infections and infestations) | 1
Varicella zoster virus infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 2
Gastrostomy failure (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Incision site oedema (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 2
Laceration (Injury, poisoning and procedural complications) | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 2
Pancreatic injury (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2
Ulna fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2
Blood creatinine increased (Investigations) | 1
Urine ketone body present (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back disorder (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chondropathy (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
SAPHO syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Insulinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Basal ganglia haemorrhage (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Complex partial seizures (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 7
Intracranial aneurysm (Nervous system disorders) | 1
Intraventricular haemorrhage (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 4
Multiple sclerosis relapse (Nervous system disorders) | 67
Optic neuritis (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 4
Status epilepticus (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 9
Tension headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Trigeminal neuralgia (Nervous system disorders) | 3
Uhthoff's phenomenon (Nervous system disorders) | 6
Abortion (Pregnancy, puerperium and perinatal conditions) | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 3
Foetal cardiac disorder (Pregnancy, puerperium and perinatal conditions) | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1
Foetal-maternal haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 1
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 1
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 1
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 2
Adjustment disorder (Psychiatric disorders) | 1
Affective disorder (Psychiatric disorders) | 1
Bipolar II disorder (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Hypomania (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 4
Post-traumatic amnestic disorder (Psychiatric disorders) | 1
Psychogenic pain disorder (Psychiatric disorders) | 1
Psychogenic tremor (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizoaffective disorder bipolar type (Psychiatric disorders) | 1
Self injurious behaviour (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 6
Suicide attempt (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Automatic bladder (Renal and urinary disorders) | 1
Calculus bladder (Renal and urinary disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Glomerulonephritis (Renal and urinary disorders) | 1
Glomerulonephritis membranous (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 4
Renal colic (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal mass (Renal and urinary disorders) | 1
Renal tubular necrosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 4
Adnexa uteri mass (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 4
Cystocele (Reproductive system and breast disorders) | 2
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 2
Menometrorrhagia (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Ovarian cyst (Reproductive system and breast disorders) | 6
Ovarian haemorrhage (Reproductive system and breast disorders) | 1
Parovarian cyst (Reproductive system and breast disorders) | 1
Pelvic adhesions (Reproductive system and breast disorders) | 1
Rectocele (Reproductive system and breast disorders) | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Vulvar dysplasia (Reproductive system and breast disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Apnoea neonatal (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Polymorphic eruption of pregnancy (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Thyroidectomy (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 4
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Pallor (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alemtuzumab (N=1314)
Tachycardia (Cardiac disorders) | 86
Autoimmune thyroiditis (Endocrine disorders) | 67
Basedow's disease (Endocrine disorders) | 165
Hyperthyroidism (Endocrine disorders) | 142
Hypothyroidism (Endocrine disorders) | 140
Vision blurred (Eye disorders) | 75
Abdominal pain (Gastrointestinal disorders) | 72
Constipation (Gastrointestinal disorders) | 104
Diarrhoea (Gastrointestinal disorders) | 170
Dyspepsia (Gastrointestinal disorders) | 71
Nausea (Gastrointestinal disorders) | 206
Vomiting (Gastrointestinal disorders) | 130
Fatigue (General disorders) | 280
Pain (General disorders) | 85
Pyrexia (General disorders) | 228
Bronchitis (Infections and infestations) | 133
Gastroenteritis (Infections and infestations) | 81
Gastroenteritis viral (Infections and infestations) | 85
Herpes zoster (Infections and infestations) | 123
Influenza (Infections and infestations) | 155
Nasopharyngitis (Infections and infestations) | 382
Oral herpes (Infections and infestations) | 78
Pharyngitis (Infections and infestations) | 68
Sinusitis (Infections and infestations) | 186
Upper respiratory tract infection (Infections and infestations) | 272
Urinary tract infection (Infections and infestations) | 360
Contusion (Injury, poisoning and procedural complications) | 141
Fall (Injury, poisoning and procedural complications) | 87
Blood creatinine increased (Investigations) | 68
Protein urine present (Investigations) | 78
Vitamin D deficiency (Metabolism and nutrition disorders) | 83
Arthralgia (Musculoskeletal and connective tissue disorders) | 216
Back pain (Musculoskeletal and connective tissue disorders) | 205
Muscle spasms (Musculoskeletal and connective tissue disorders) | 132
Muscular weakness (Musculoskeletal and connective tissue disorders) | 113
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 75
Myalgia (Musculoskeletal and connective tissue disorders) | 80
Pain in extremity (Musculoskeletal and connective tissue disorders) | 189
Dizziness (Nervous system disorders) | 130
Headache (Nervous system disorders) | 437
Hypoaesthesia (Nervous system disorders) | 176
Multiple sclerosis (Nervous system disorders) | 70
Multiple sclerosis relapse (Nervous system disorders) | 508
Paraesthesia (Nervous system disorders) | 168
Anxiety (Psychiatric disorders) | 133
Depression (Psychiatric disorders) | 154
Insomnia (Psychiatric disorders) | 231
Haematuria (Renal and urinary disorders) | 92
Proteinuria (Renal and urinary disorders) | 122
Cough (Respiratory, thoracic and mediastinal disorders) | 127
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 91
Rash (Skin and subcutaneous tissue disorders) | 208
Rash generalised (Skin and subcutaneous tissue disorders) | 110
Urticaria (Skin and subcutaneous tissue disorders) | 96
Flushing (Vascular disorders) | 79
Hypertension (Vascular disorders) | 92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.